CLINICAL TRIAL: NCT02848391
Title: Impact of Hypobaric Flight Simulation on Walking Endurance in COPD Patients
Brief Title: Hypobaric Flight Simulation in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Kloster Grafschaft (Other)
Responsible Party: Principal Investigator, Dominic Dellweg, M.D., PD Dr. med, Krankenhaus Kloster Grafschaft
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Airtravel01
Record Dates: First submitted 2016-06-24; First posted 2016-07-28 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: COPD; Hypoxia; Aviation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia | interventions — Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy subjects (Experimental): three hour flight simulation
  Interventions: Other: Environmental
- COPD normocapnic (Experimental): three hour flight simulation
  Interventions: Other: Environmental
- COPD hypercapnic (Experimental): three hour flight simulation
  Interventions: Other: Environmental

INTERVENTIONS:
Other: Environmental — hypobaric flight simulation

SUMMARY:
Aim of this study was to evaluate the hypoxic response during hypobaric flight simulation in normal individuals as well as in normocapnic and hypercapnic COPD patients as well as to evaluate the impact of a flight simulation on walking endurance in these patients.

DETAILED DESCRIPTION:
Background and aim:

Commercial aircrafts have their altitude compensation adjusted to 2500 meter above sea level which corresponds to a pressure difference of about 270 hPa. This causes a reduction of the partial pressure of oxygen during the flight. Patients with lung disease are especially challenged by large walking distances within airports and during their journey. The objective of our study is to evaluate the impact of a simulated flight under hyperbaric conditions on walking endurance in healthy individuals as well as in COPD Patients with and without hypercapnia.

Method:

Healthy individuals as well as COPD patients were assessed pre-flight with the following measurements:

1. Arterial blood gas analysis
2. Lung function test
3. Lung diffusion test
4. Hemoglobin level
5. Six minute walking distance

During the flight measurements included (measured every 30 minutes until landing):

1. Heartrate
2. Oxygen saturation
3. Borg scale

Post flight measurements included:

1. Arterial blood gas analysis
2. Six minute walking distance

Intended analysis:

* Description of endurance response as a function of COPD disease severity.
* Description of endurance response in normocapnic and hypercapnic COPD patients.
* Detection of pre-flight predictors that determine flight tolerability and hypoxic response.

ELIGIBILITY:
Inclusion Criteria:

* No lung disease
* COPD without hypercapnea
* COPD with hypercapnea

Exclusion Criteria:

* Claustrophobia
* Renal insufficiency
* Heart failure (ejection fraction < 45 %)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in six minute walking distance measured in meters | 30 Minutes before and after a 3 hour simulated flight (Time point - 30 and + 210 minutes)
  difference between pre- and post-flight walking distance

SECONDARY OUTCOMES:
minimal Oxygen saturation measured by pulse oxymetry in % | measurement completed at 180 minutes
  Nadir of the oxygen saturation during the flight

CONTACTS AND LOCATIONS:
Locations (1):
- Kloster Grafschaft, Schmallenberg, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No